CLINICAL TRIAL: NCT01265953
Title: Chemoprevention of Prostate Cancer, HDAC Inhibition and DNA Methylation
Acronym: PBroC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon State University (Other); OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Jackilen Shannon, Staff Scientist, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Portland VA-09-0607; 2096 (Other: PVAMC IRB); 6232 (Other: OHSU IRB); 2P01CA090890-06A2 (NIH)
Record Dates: First submitted 2010-12-16; First posted 2010-12-23 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer Prevention
Keywords: cancer prevention; isothiocyanate; sulforaphane
MeSH Terms: interventions — sulforaphane; Gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SFN-rich broccoli sprout extract capsules (Experimental): Four weeks SFN-rich broccoli sprout extract (BSE) capsules: 200µmol of sulforaphane (SFN) daily, 2 capsules (1 capsule B.I.D.) daily
  Interventions: Drug: SFN-rich broccoli sprout extract capsules
- Placebo capsules (Placebo Comparator): Four weeks placebo capsules: 2 capsules (1 capsule B.I.D.) daily
  Interventions: Dietary Supplement: Gelatin capsule containing microcrystalline cellulose.

INTERVENTIONS:
Drug: SFN-rich broccoli sprout extract capsules — Four weeks SFN-rich broccoli sprout extract (BSE) capsules: 200µmol of SFN, 2 capsules (1 capsule B.I.D.) daily
  Other Names: BSE; SFN; Sulforaphane
  Arms: SFN-rich broccoli sprout extract capsules
Dietary Supplement: Gelatin capsule containing microcrystalline cellulose. — Four weeks placebo capsules: 2 capsules (1 capsule B.I.D.) daily
  Arms: Placebo capsules

SUMMARY:
The objective of the study is to identify mechanisms by which compounds found in cruciferous vegetables alter gene expression via epigenetic modifications (changes in gene expression) and may prevent prostate cancer development.

The investigators have found that sulforaphane (SFN), an isothiocyanate found in cruciferous vegetables, inhibits histone deacetylase (HDAC) activity in human colorectal and prostate cancer cells.

DETAILED DESCRIPTION:
Prostate cancer is the most frequently diagnosed non-cutaneous cancer and is the second leading cause of cancer death in American men. The precise etiologic factors that initiate and enhance the progression of prostate cancer remain unknown, but epigenetic alterations and diet/lifestyle factors have come forth as significant contributing factors. Epidemiologic studies suggest that cruciferous vegetable intake decreases the risk for prostate cancer. The long-term goal of this proposal is to identify mechanisms by which dietary compounds, such as those found in cruciferous vegetables decrease prostate cancer risk. The objective of the study is to identify mechanisms by which compounds found in cruciferous vegetables alter gene expression via epigenetic modifications and may prevent prostate cancer development.

The investigators have found that SFN, an isothiocyanate found in cruciferous vegetables, inhibits HDAC activity in human colorectal and prostate cancer cells.

Targeting the epigenome, including the use of HDAC and DNA methyltransferase (DNMT) inhibitors, is an evolving strategy for cancer chemoprevention and both have shown promise in cancer clinical trials.

This Randomized, Double Blind, Clinical Trial will address the following objectives:

1. Identify distribution of SFN and its metabolites and HDAC inhibition following supplementation with an SFN-rich broccoli sprout extract in subjects at risk for prostate cancer (Primary Endpoints)
2. Investigate the effects of supplementation with an SFN-rich broccoli sprout extract on DNA methylation status and proliferation markers in a pre-biopsy setting (secondary analysis)

The effects of short-term supplementation with an SFN-rich broccoli sprout extract on benign epithelial tissue will be studied in men characterized as being at risk for prostate cancer in a randomized, placebo-controlled trial. Men scheduled for prostate biopsy will be recruited into the trial.

Following successful completion of the consent, two 10 mL blood specimens for study analyses, a 4 mL specimen for total bilirubin assessment will be drawn and the subject will provide a urine sample. The study coordinator will explain the Diet History questionnaires (DHQ) and administer the risk factor and adverse event (AE) questionnaires in order to obtain data on potential confounding dietary variables and gain subjects' baseline symptoms.

The study coordinator will provide the subject with a month' supply of either an SFN-rich broccoli sprout extract (BSE) capsule which consist of 200µmol of sulforaphane (SFN) or matching placebo, as dispensed by the Research Pharmacy. The matching placebo for the BSE consists of a gelatin capsule containing microcrystalline cellulose.

Around every 2 weeks, study coordinator will call to complete AE reporting and any changes in medications or supplements and complete brief cruciferous vegetable intake checklist. Subjects will return any unused study "drug" to the study coordinator at the time of biopsy (or at the 4 week visit if subject's prostate biopsy is delayed).

ELIGIBILITY:
Inclusion Criteria:

* Men scheduled for a prostate biopsy
* Age 21 years or older
* Signed informed subject consent

Exclusion Criteria:

* Definitive diagnosis with prostate cancer
* Significant active medical illness which in the opinion of the investigator or clinician would preclude protocol treatment
* Diagnosis of liver disease as noted on the patient problem list or baseline total bilirubin greater than institutional upper limit of normal
* Subject reported allergy or sensitivity to cruciferous vegetables
* Use of oral antibiotics, with the exception of doxycycline, within three months prior to randomization
* Use of warfarin or need for therapeutic anticoagulation at time of biopsy or at anytime during the course of the trial.
* Current oral steroid therapy
* Current therapy with valproate or other pharmacological drugs associated with HDAC inhibition
* Diagnosed dementia as noted on the patient problem list or other significant mental illness that may impact the subjects' ability to follow instructions or comply with the study protocol
* Patient may not be a part of another flagged study
* Patients already taking SFN dietary supplements

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jackilen Shannon, PhD, Principal Investigator — Portland VA Medical Center
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon

REFERENCES:
- [Derived] Zhang Z, Garzotto M, Davis EW 2nd, Mori M, Stoller WA, Farris PE, Wong CP, Beaver LM, Thomas GV, Williams DE, Dashwood RH, Hendrix DA, Ho E, Shannon J. Sulforaphane Bioavailability and Chemopreventive Activity in Men Presenting for Biopsy of the Prostate Gland: A Randomized Controlled Trial. Nutr Cancer. 2020;72(1):74-87. doi: 10.1080/01635581.2019.1619783. Epub 2019 Jun 1. PMID 31155953

RESULTS

PARTICIPANT FLOW:
Groups:
- Supplement: Subjects in this group were administered with broccoli sprout extract.
- Placebo: Subjects in this group were administered with placebo.
Period: Overall Study
Arm/Group | Supplement | Placebo
Started | 50 | 48
Completed | 45 | 45
Not Completed | 5 | 3
Not completed — Non compliance | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Broccoli Sprout Extract Capsules: Four weeks broccoli sprout extract (BSE) capsules: 200µmol of sulforaphane (SFN) daily, 2 capsules (1 capsule B.I.D.) daily
- Placebo Capsules: Four weeks placebo capsules: 2 capsules (1 capsule B.I.D.) daily
  Dietary Supplement: Gelatin capsule containing microcrystalline cellulose
- Total: Total of all reporting groups
Arm/Group | Broccoli Sprout Extract Capsules | Placebo Capsules | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (5.4) | 64.9 (5.0) | 65.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 48 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 48 | 46 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 48 | 98
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (7.6) | 31.1 (6.4) | 30.0 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Change of Total Urine SFN (Sulforaphane) Metabolites
Description: Collection of blood and urine specimens occurred at pre-intervention and post-intervention. Change = post-intervention level minus pre-intervention level
Time Frame: Baseline and 4-8 weeks following intervention
Population: Not all subjects had urine samples for analysis, therefore, the total number of subjects in this urine analysis is different from total number of enrolled subjects.
Measure: Mean (Standard Error); unit: micromolar (µM) concentrations of urina
Arm/Group | Supplement | Placebo
Number analyzed (Participants) | 42 | 44
micromolar (µM) concentrations of urina | 4.75 (0.64) | -0.02 (0.01)

2. Primary Outcome: Change of Total Plasma SFN (Sulforaphane) Metabolites Level
Description: In subjects at risk for prostate cancer, presence of SFN was analyzed in plasma. Collection of blood specimens occurred at pre-intervention and post-intervention. The Change = post-intervention level minus pre-intervention level
Time Frame: Baseline and 4-8 weeks following intervention
Population: We missed blood samples from some subjects, therefore, total number of subjects analyzed for the plasma-based analysis is different from the number of total enrolled subjects.
Measure: Mean (Standard Error); unit: micromolar (µM)
Arm/Group | Supplement | Placebo
Number analyzed (Participants) | 42 | 44
micromolar (µM) | 0.12 (0.03) | -0.0003 (0.0002)

3. Primary Outcome: Percentage of Ki67 Positive Cells up to 8 Weeks Post-randomization
Description: Ki67 is a biomarker of disease progression. Immunohistochemical (IHC) analysis of Ki67 was performed using research only prostate biopsy specimens collected post-intervention at the time of the clinically-indicated prostate biopsy.
Time Frame: Baseline and 4-8 weeks following intervention; prostate biopsy were collected post-intervention when clinically-indicated
Population: Some subjects did not have post-intervention prostate tissue that can be used for IHC analysis, therefore, the overall number of participants analyzed for IHC analysis is different from the total enrolled subjects.
Measure: Mean (Standard Error); unit: percent positive
Arm/Group | Supplement | Placebo
Number analyzed (Participants) | 41 | 42
percent positive | 1.8 (0.2) | 1.9 (0.3)

4. Primary Outcome: Expression of Histone Deacetylase 6 (HDAC6)
Description: Immunohistochemical (IHC) analysis of HDAC6 expression using research-only prostate biopsy tissue collected post-intervention at the time of the clinically-indicated prostate biopsy. A modified Histo-score (H-score) was calculated, which involved semiquantitative assessment of both staining intensity (graded as 1-3 with 1 representing weak staining, 2 moderate, and 3 strong) and percentage of positive cells. H-score ranged from 0 to 300 with 300 the strongest expression.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Error); unit: H-score
Arm/Group | Supplement | Placebo
Number analyzed (Participants) | 41 | 42
H-score | 187 (13) | 183 (12.5)

ADVERSE EVENTS:
Arm/Group | Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/48
Other Adverse Events (participants affected / at risk) | 2/50 | 1/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supplement (N=50) | Placebo (N=48)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Taste Alteration (Nervous system disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No